CLINICAL TRIAL: NCT02203981
Title: TopQ Cut-off Determination Study For 3D-OCT 1 Maestro and 3D OCT-2000
Status: Completed | Type: Observational
Sponsor: Topcon Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Organization: Topcon Corporation (Industry)
Other Study IDs: TopQ_Maestro_OCT2000_001
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Healthy
Keywords: normal Eyes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To determine optimal cut-off value for the TopQ cut-off on the Maestro and 3D OCT-2000.

ELIGIBILITY:
Inclusion Criteria:

* No known ocular pathologies

Exclusion Criteria:

* Any known ocular pathologies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects that have no known ocular pathologies
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2014-01; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Retinal Thickness | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Sunni Patel, PhD, Principal Investigator — Topcon Corporation
Locations (1):
- Topcon Medical Systems, Inc., Oakland, New Jersey, United States